CLINICAL TRIAL: NCT02701374
Title: TRK-700 An Early Phase II Study in Patients With Post-Herpetic Neuralgia -Double Blind Comparison With Placebo-
Brief Title: Efficacy and Safety of TRK-700 in Patient With Post-Herpetic Neuralgia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Toray Industries, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 700PNC01
Record Dates: First submitted 2016-02-26; First posted 2016-03-08 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Post-Herpetic Neuralgia
Keywords: TRK-700; Post-Herpetic Neuralgia
MeSH Terms: conditions — Neuralgia, Postherpetic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1:TRK-700 (Experimental): high dose
  Interventions: Drug: TRK-700
- 2:TRK-700 (Experimental): low dose
  Interventions: Drug: TRK-700
- 3:Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TRK-700
  Arms: 1:TRK-700; 2:TRK-700
Drug: Placebo
  Arms: 3:Placebo

SUMMARY:
In Post-Herpetic Neuralgia(PHN) patients:

* To conduct an explorative investigation of the efficacy and safety of repeated oral doses of TRK-700 via a randomized double blind comparative study
* To measure the plasma concentration of TRK-700 and its metabolites

ELIGIBILITY:
Inclusion Criteria:

* Patients with pain persisting for at least 3 months after the onset of herpes zoster
* Patients whose average pain score on the Numerical Rating Scale (NRS) over the past 24 hours at preliminary enrollment is at least 4

Exclusion Criteria:

* Patients with another skin disease that may affect the evaluation of the pain at the site of PHN
* Patients with pain other than PHN that may affect the evaluation of pain
* Patients with pain that is suspected to be mainly psychogenic
* Patients who have received neurolytic or neurosurgical therapy for PHN

Ages: 20 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2016-03; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Change in average Numerical Rating Scale (NRS) | baseline to week 8
  Change in average NRS collected by Pain Diary from baseline to week 8 in subjects receiving TRK-700 versus Placebo

CONTACTS AND LOCATIONS:
Locations (1):
- Tokyo, Tokyo, Japan